CLINICAL TRIAL: NCT06737198
Title: Correlation of Preoperative Indices (serum Vit D, Calcium, Phosphorus, FAR, PLR, SII) on Intraoperative Bleeding in CRS
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20241112-07
Record Dates: First submitted 2024-12-03; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinosinusitis (CRS) with and Without Nasal Polyps
Keywords: chronic rhinosinusitis; Intraoperative haemorrhage
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- chronic rhinosinusitis: chronic rhinosinusitis with/without nasal polys.
  Interventions: Other: without interventios.

INTERVENTIONS:
Other: without interventios. — without interventios.

SUMMARY:
The purpose of this observational study was to examine whether preoperative indicators correlate with intraoperative bleeding to facilitate control of intraoperative bleeding.

DETAILED DESCRIPTION:
In this study, we analysed the effect of preoperative inflammation on intraoperative haemorrhage at the subjective and objective levels by measuring a number of indicators (including Vit D, Ca, P, and some ratios) in the blood specimens and by three scales.Blood test indicators can be obtained from routine tests.Three scales were obtained by the researcher after interviewing the patients, Symptom Score (0-15), where higher scores indicate more severe symptoms, Lund-Kennedy Score (0-6), where higher scores indicate higher levels of localised inflammation, Lund-Mackay Score (0-12 unilaterally and 24 bilaterally), where higher scores indicate higher levels of inflammation, and Lund-Mackay Score (0-12 unilaterally and 24 bilaterally), where higher scores indicate higher levels of inflammation.Lund-Mackay score (0-12 unilaterally, 24 bilaterally), where higher scores represent higher levels of inflammation.Final correlation of blood test indices and three scale scores with intraoperative.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic rhinosinusitis

Exclusion Criteria:

Sinus cyst Upper respiratory tract infection in the last 1 week Use of antiepileptic drugs Use of aspirin Use of anticoagulant or antiplatelet drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with chronic sinusitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative haemorrhage | 2024/11/1-2025/7/31
  Intraoperative haemorrhage was grouped with a cut-off value of 150 ml and divided into <150 ml (normal haemorrhage group) and ≥150 ml (high haemorrhage group).

SECONDARY OUTCOMES:
Symptom system | 2024/11/1-2025/7/31
  Symptom system (0-15 scores), assessed in five areas: nasal congestion, runny nose, reduced sense of smell, head and face swelling, and sleep disturbances, where higher scores represent more severe symptoms.
Lund-Kennedy system | 2024/11/1-2025/7/31
  Lund-Kennedy system (0-6 scores), assessed under nasal endoscopy in terms of polyps, oedema and nasal secretions, where a higher score represents a higher level of local inflammation.
Lund-Mackay system | 2024/11/1-2025/7/31
  The Lund-Mackay system (0-12 unilaterally, 24 points in total bilaterally) analyses the inflammatory status within each sinus and the assessment of whether the sinonasal complex is obstructed in two major ways, where higher scores represent higher levels of inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No